CLINICAL TRIAL: NCT00404417
Title: Botulinum Toxin A for the Treatment of Chronic Lumbar Back Pain: A Prospective Randomized Double-blind Placebo-controlled Crossover Study
Brief Title: Botulinum Toxin A for the Treatment of Chronic Lumbar Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: COL (ret) Kevin R. Cannard, MD, Walter Reed Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DCI P06-71038
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Low Back Pain
Keywords: pain; lumbar
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Botox/Placebo
  Interventions: Drug: Botulinum Toxin A / Placebo
- 2 (Experimental): Botox/Botox
  Interventions: Drug: Botulinum Toxin A / Botulinum Toxin A
- 3 (Experimental): Placebo/Botox
  Interventions: Drug: Placebo / Botulinum Toxin A
- 4 (Placebo Comparator): Placebo/Placebo
  Interventions: Drug: Placebo / Placebo

INTERVENTIONS:
Drug: Botulinum Toxin A / Placebo — Botulinum Toxin A at first injection / Placebo at second injection
  Other Names: Botox
  Arms: 1
Drug: Botulinum Toxin A / Botulinum Toxin A — Botulinum Toxin A at first injection / Botulinum Toxin A at second injection
  Other Names: Botox
  Arms: 2
Drug: Placebo / Botulinum Toxin A — Placebo at first injection / Botulinum Toxin A at second injection
  Other Names: Botox
  Arms: 3
Drug: Placebo / Placebo — Placebo at first injection / Placebo at second injection
  Other Names: Placebo
  Arms: 4

SUMMARY:
This study will assess the efficacy and the duration of efficacy of Botulinum toxin A (Botox®) injected into the lumbar paraspinal muscles for reducing pain and disability in subjects suffering from chronic low back pain of six months duration or longer and arising from an identifiable muscle strain injury or back trauma. The treatment modality and techniques used are based on a successful prior 4 month open-labeled pilot study done by this research group, but will employ a prospective double-blind, randomized, cross-over design to control for any placebo or mechanical trigger-point injection effects. Subjects will also be assessed for a longer duration to better define the duration of efficacy.

DETAILED DESCRIPTION:
One hundred sixty subjects will be randomly assigned to one of four arms (placebo/placebo, placebo/Botox, Botox/placebo, Botox/Botox). In the first of two phases, randomized subjects will blindly receive either Botox® (study arms Botox/placebo and Botox/Botox) or placebo (study arms placebo/placebo and placebo/Botox) injection into the lumbar paraspinal muscles. The subjects will be assessed using validated scales for pain and disability prior to injection and monthly thereafter for four months. In the second phase, a second set of lumbar injections will be administered based on the initial randomization and will blindly receive either Botox® (study arms placebo/Botox and Botox/Botox) or placebo (study arms placebo/placebo and Botox/placebo) injection into the lumbar paraspinal muscles. The subjects will again be assessed using the same validated scales for pain and disability, prior to injection and monthly thereafter, but for six months to extend the monitoring period to better define the limits of duration of effect.

This will result in half of the subjects being crossed-over from Botox® to placebo (study arm Botox/placebo) or vice versa (study arm placebo/Botox) and one quarter of subjects receiving two courses of either Botox® alone (Botox/Botox) or placebo alone (placebo/placebo). All subjects will continue to receive medication and/or physiotherapy per standard of care but those treatments will be recorded and controlled for in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military, retired military or other DoD healthcare beneficiaries of either sex, aged 18-70 years, with symptoms of chronic back pain.
* A clear history of an identifiable muscle strain or back trauma preceding the chronic pain.
* Current pain duration > 6 months.
* MRI of the affected spine area to define potential or serious pathology as per standard of care.
* Written informed consent and written authorization for use or release of health and research study information.
* Normal neurological examination without evidence of radiculopathy.
* VAS score minimum of 4 cm or reaches an average of 4 cm out of 10 cm at least 4 days a week, at time of entry into study
* Ability to follow study instructions and likely to complete all required visits.
* Negative urine pregnancy test prior to the administration of study medication (for females of childbearing potential) (if applicable).

Exclusion Criteria:

* Age less than 18 or greater than 70 years
* Concomitant use of amino glycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
* Any medical condition that may put the subject at increased risk with exposure to Botulinum Toxin A (Botox®), including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis/motor neuron disease, neuropathy, renal stones, or any other disorder that might interfere with neuromuscular function or produce a similar type of back pain.
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Known allergy or sensitivity to any of the components in the study medication.
* Evidence of recent alcohol or substance abuse.
* Known, uncontrolled systemic disease.
* Participation in the 30 days preceding enrollment or during the duration of this study in another investigational drug or device study.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Significant Axis I or Axis II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into study
* Duration of back pain < 6 months.
* Thoracic or cervical spine pain in the absence of low back pain.
* Anesthetic or corticosteroid injection to the lumbosacral spine within 8 weeks of enrollment.
* Any anesthetic or steroid injections into any back muscles in the 4 weeks prior to enrollment.
* A prior spine MRI or CT (any region) with evidence of significant pathology of the spinal cord, roots, or elements of the spinal column to include; impingement on the spinal cord or nerve roots, intrinsic pathology of the spinal cord (e.g. syrinx) or nerve roots, evidence of a neoplastic or infectious process involving the spinal cord or nerve roots or structural elements of the spine (e.g. vertebra or intervertebral disks), or any deformities of the bony or supporting elements of the spinal column that deform the spinal cord or the nerve roots. Nonspecific degenerative changes of the spine, Schmorl's nodules, and other similar findings that do not impinge upon or involve the spinal cord or nerve roots will not be considered exclusionary.
* Signs of radiculopathy on neurological examination.
* History of back surgery within one year or incomplete resolution of back pain due to a previous surgery (persistence of back pain present prior to surgery, i.e. a surgical failed back, is not exclusionary).
* Subjects involved in litigation, seeking significant disability for low back pain, or with evident secondary gain as determined by the neurologist through chart review and patient interview.
* Any previous use of Botox®, Dysport® or Myobloc®. Previous use of Botox Cosmetic or Myobloc for cosmetic purposes is allowed if the last administration occurred over 6 months prior to enrollment and the injected dose was less than or equal to 30 units (or an equivalent dose of Myobloc). Copies of all records of Botox Cosmetic or Myobloc injection(s) must be provided by the subject prior to enrollment for verification.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
relief of chronic low back pain | 8 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Cannard, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Pope MH, Frymoyer JW, Krag MH. Diagnosing instability. Clin Orthop Relat Res. 1992 Jun;(279):60-7. PMID 1600673
- [Background] Wipf JE, Deyo RA. Low back pain. Med Clin North Am. 1995 Mar;79(2):231-46. doi: 10.1016/s0025-7125(16)30065-7. PMID 7877388
- [Background] Cherkin DC, Sherman KJ, Deyo RA, Shekelle PG. A review of the evidence for the effectiveness, safety, and cost of acupuncture, massage therapy, and spinal manipulation for back pain. Ann Intern Med. 2003 Jun 3;138(11):898-906. doi: 10.7326/0003-4819-138-11-200306030-00011. PMID 12779300
- [Background] Grazko MA, Polo KB, Jabbari B. Botulinum toxin A for spasticity, muscle spasms, and rigidity. Neurology. 1995 Apr;45(4):712-7. doi: 10.1212/wnl.45.4.712. PMID 7723960
- [Background] Aoki KR. Pharmacology and immunology of botulinum toxin serotypes. J Neurol. 2001 Apr;248 Suppl 1:3-10. doi: 10.1007/pl00007816. PMID 11357237